CLINICAL TRIAL: NCT00819988
Title: A Randomized, Double-blind, Placebo-controlled Trial to Assess the Safety and Efficacy of the Perioperative Administration of Pregabalin in Reducing the Incidence of Postoperative Delirium and Improving Acute Postoperative Pain Management
Brief Title: Pregabalin in the Prevention of Postoperative Delirium and Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Dr. A. Chaput, Clinician Investigator, Ottawa Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PSI2008525
Record Dates: First submitted 2009-01-08; First posted 2009-01-09 (Estimated); Last update posted 2012-01-10 (Estimated); Status verified 2012-01

CONDITIONS: Delirium; Pain
Keywords: Postoperative; Perioperative; Orthopedic surgery; Vascular surgery; Gabapentinoid
MeSH Terms: conditions — Delirium; Pain | interventions — Pregabalin; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugar pill (Placebo Comparator): Single dose given 30-60 minutes preoperatively, then given every 8 hours for 3 days postoperatively
  Interventions: Other: Sugar pill
- Pregabalin (Experimental): Single dose of 75 mg given 30-60 minutes preoperatively, then 50 mg every 8 hours for 3 days postoperatively if creatinine clearance > 60 ml/min OR 25 mg every 8 hours for 3 days postoperatively if creatinine clearance 30-60 ml/min
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Pregabalin — Pregabalin capsule 75 mg given preoperatively, then eith 50 mg or 25 mg given every 8 hours for 3 days postoperatively based on renal function
  Other Names: Lyrica
  Arms: Pregabalin
Other: Sugar pill — Single dose given 30-60 minutes preoperatively, then given every 8 hours for 3 days postoperatively
  Arms: Sugar pill

SUMMARY:
The purpose of this study is to determine whether administration of pregabalin by mouth immediately preoperatively and three times daily for 3 days after surgery reduces the incidence of delirium postoperatively and improves overall pain control.

DETAILED DESCRIPTION:
Delirium is a common postoperative complication occurring in up to 73% of patients sometime during their hospital stay. Elderly patients undergoing major surgical procedures are at highest risk. While many risk factors for delirium are known, the specific pathophysiology of postoperative delirium remains unclear and is likely multifactorial. The most common inciting agents and events include metabolic causes, medications, blood loss, hypoxemia and pain. Pain and its management are intimately related to the likelihood of developing postoperative delirium. As a class, gabapentinoids, such as pregabalin, have proven to reduce postoperative pain and narcotic consumption and therefore may have a role to play in the prevention of postoperative delirium.

ELIGIBILITY:
Inclusion Criteria:

* aged 60 years and older
* booked for major orthopaedic or vascular procedure
* expected length of stay > 2 days

Exclusion Criteria:

* open AAA repair
* EVAR
* allergy/sensitivity to pregabalin or gabapentin
* use of pregabalin or gabapentin in previous 14 days
* severe liver disease
* severe renal dysfunction defined as either having creatinine clearance < 30 ml/min or being dialysis-dependent
* seizure disorder
* MMSE < 24/30
* inability to speak English or French

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2009-05; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Delirium (patient is either CAM-ICU positive or positive for delirium by chart review) | postoperative day 1, 2, 3

SECONDARY OUTCOMES:
Interference with daily activities using BPI | postoperative day 3
Pain at rest using NRS | postoperative days 1, 2, 3
Pain with movement of the operative site using NRS | postoperative days 1, 2, 3
Narcotic analgesic requirements | postoperative days 0, 1, 2, 3
Sedation using RSS | postoperative days 1, 2, 3
Narcotic-related adverse effects using ORSDS | postoperative days 1, 2, 3
Recovery using the QoR | postoperative day 3
Length of stay | Discharge day
Medical Outcome Study (MOS) sleep score | Postoperative day 3

CONTACTS AND LOCATIONS:
Overall Officials: Alan J Chaput, MD, MSc, Principal Investigator — The Ottawa Hospital; Homer Yang, MD, Study Director — The Ottawa Hospital; Gregory L Bryson, MD, MSc, Study Director — The Ottawa Hospital; Holly Evans, MD, Study Director — The Ottawa Hospital; Paul Beaule, MD, Study Director — The Ottawa Hospital; Prasad Jetty, MD, Study Director — The Ottawa Hospital; Barbara Power, MD, Study Director — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Inouye SK, van Dyck CH, Alessi CA, Balkin S, Siegal AP, Horwitz RI. Clarifying confusion: the confusion assessment method. A new method for detection of delirium. Ann Intern Med. 1990 Dec 15;113(12):941-8. doi: 10.7326/0003-4819-113-12-941. PMID 2240918
- [Background] Bitsch M, Foss N, Kristensen B, Kehlet H. Pathogenesis of and management strategies for postoperative delirium after hip fracture: a review. Acta Orthop Scand. 2004 Aug;75(4):378-89. doi: 10.1080/00016470410001123. PMID 15370579
- [Background] Morrison RS, Magaziner J, Gilbert M, Koval KJ, McLaughlin MA, Orosz G, Strauss E, Siu AL. Relationship between pain and opioid analgesics on the development of delirium following hip fracture. J Gerontol A Biol Sci Med Sci. 2003 Jan;58(1):76-81. doi: 10.1093/gerona/58.1.m76. PMID 12560416
- [Background] Bekker AY, Weeks EJ. Cognitive function after anaesthesia in the elderly. Best Pract Res Clin Anaesthesiol. 2003 Jun;17(2):259-72. doi: 10.1016/s1521-6896(03)00005-3. PMID 12817919
- [Background] Lynch EP, Lazor MA, Gellis JE, Orav J, Goldman L, Marcantonio ER. The impact of postoperative pain on the development of postoperative delirium. Anesth Analg. 1998 Apr;86(4):781-5. doi: 10.1097/00000539-199804000-00019. PMID 9539601
- [Background] Gilron I. Review article: the role of anticonvulsant drugs in postoperative pain management: a bench-to-bedside perspective. Can J Anaesth. 2006 Jun;53(6):562-71. doi: 10.1007/BF03021846. PMID 16738290
- [Background] Peng PW, Wijeysundera DN, Li CC. Use of gabapentin for perioperative pain control -- a meta-analysis. Pain Res Manag. 2007 Summer;12(2):85-92. doi: 10.1155/2007/840572. PMID 17505569
- [Background] Leung JM, Sands LP, Rico M, Petersen KL, Rowbotham MC, Dahl JB, Ames C, Chou D, Weinstein P. Pilot clinical trial of gabapentin to decrease postoperative delirium in older patients. Neurology. 2006 Oct 10;67(7):1251-3. doi: 10.1212/01.wnl.0000233831.87781.a9. Epub 2006 Aug 16. PMID 16914695